CLINICAL TRIAL: NCT02643771
Title: Clinical and Microbiological Evaluation of Non-surgical Periodontal Treatment of Diabetic and Non-diabetic Patients: A Longitudinal Study
Brief Title: Clinical and Microbiological Evaluation of Periodontal Treatment of Diabetic Patients: A Longitudinal Study
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Eduardo Aleixo Figueira (Other)
Collaborators: Coordenação de Aperfeiçoamento de Pessoal de Nível Superior. (Other Government)
Responsible Party: Sponsor-Investigator, Eduardo Aleixo Figueira, DDS, MSc, PhD, Post-Doctoral Student, Universidade Federal do Rio Grande do Norte
Organization: Universidade Federal do Rio Grande do Norte (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: U1111-1175-5481
Record Dates: First submitted 2015-12-28; First posted 2015-12-31 (Estimated); Last update posted 2015-12-31 (Estimated); Status verified 2015-12

CONDITIONS: Chronic Periodontitis; Diabetes Mellitus, Type 2
Keywords: Dental Scaling; Blood Glucose; Hemoglobin A, Glycosylated
MeSH Terms: conditions — Chronic Periodontitis; Diabetes Mellitus, Type 2 | interventions — Root Planing

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Diabetic group (Experimental): Subjects with Chronic Periodontitis and Type 2 Diabetes Mellitus treated with non surgical periodontal therapy (Full Mouth Scaling and Root Planing)
  Interventions: Procedure: Full Mouth Scaling and Root Planing
- Nondiabetic group (Experimental): Subjects with Chronic Periodontitis and without Type 2 Diabetes Mellitus treated with non surgical periodontal therapy (Full Mouth Scaling and Root Planing)
  Interventions: Procedure: Full Mouth Scaling and Root Planing

INTERVENTIONS:
Procedure: Full Mouth Scaling and Root Planing — This procedure was performed as described by Quirynen et al. 2005 with some modifications

SUMMARY:
The purpose of this study is to determine whether periodontal treatment improves the periodontal clinical parameters in the periodontal patients with diabetes regarding non-diabetics: two years follow-up.

DETAILED DESCRIPTION:
All the subjects in the study will receive non surgical periodontal treatment in one session (full-mouth scaling and root planing). Clinical parameters will be assessed in all teeth (except third molars) by one experienced and trained examiner before treatment and every 3 months for 2 years. Visible plaque index (VPI) will be represented a mean percentage of sites with visible plaque calculated for all teeth analyzed (four sites per tooth). Others parameters will be assessed at six sites per tooth using a manual periodontal probe (15mm). Bleeding on probing (BOP) will be represented the mean percentage of sites with bleeding (up to 15 seconds after probing) calculated for all teeth analyzed. Probing depth (PD - distance between the gingival margin and the bottom of the sulcus/pocket), gingival recession (GR - distance between the cementoenamel junction and gingival margin) and clinical attachment level (CAL - distance between the cementoenamel junction and the bottom of the sulcus/pocket) will be represented a mean distance calculated per site for all teeth analyzed. For blood parameters, an outside laboratory will perform all blood analysis. It will be requested for each subject with diabetes (DG) at baseline, each 3 months post-treatment. Fasting plasma glucose (FPG) will be expressed in milligrams per deciliter and HbA1c will be expressed as a percentage. Statistical analysis will be performed using an available software program and the patient will be considered as the unit of analysis.The data will be processed and analyzed by descriptive and inferential statistics, probably nonparametric.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of chronical periodontitis according to Lopez et al. 2002 (one or more teeth with at least one site with PD >= 4mm or CAL >= 3mm);
* And have at least 8 natural teeth (excluding third molars), and older than 18 years and of both genders.

Exclusion Criteria:

* Any systemic diseases or complications (except Type 2 Diabetes Mellitus) such as cardiovascular disease, Alzheimer's, lung or brain diseases and metabolic syndrome;
* Use of antibiotics or periodontal treatment within the past 6 months;
* Long-term administration of anti-inflammatory or/and immunosuppressive agents;
* Current smoker or former smoker for the past 5 years;
* Pregnant or breastfeeding;
* And presence of orthodontic appliances.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 144 (Estimated)
Dates: Start 2013-01; Primary Completion 2016-10 (Estimated); Study Completion 2017-10 (Estimated)

PRIMARY OUTCOMES:
Percentage of bleeding on probing | Baseline
  The mean percentage of periodontal sites with bleeding on probing
Percentage of bleeding on probing | at three months
  The mean percentage of periodontal sites with bleeding on probing
Percentage of bleeding on probing | at six months
  The mean percentage of periodontal sites with bleeding on probing
Percentage of bleeding on probing | at nine months
  The mean percentage of periodontal sites with bleeding on probing
Percentage of bleeding on probing | at twelve months
  The mean percentage of periodontal sites with bleeding on probing
Percentage of bleeding on probing | at eighteen months
  The mean percentage of periodontal sites with bleeding on probing
Percentage of bleeding on probing | at twenty four months
  The mean percentage of periodontal sites with bleeding on probing

SECONDARY OUTCOMES:
Percentage of visible plaque index | Baseline and at three, six, nine, twelve, eighteen and twenty four months
  The mean percentage of periodontal sites with visible plaque
Probing depth (mm) | Baseline and at three, six, nine, twelve, eighteen and twenty four months
  The mean of probing depth in millimeters calculated for periodontal sites.
Clinical attachment level (mm) | Baseline and at three, six, nine, twelve, eighteen and twenty four months
  The mean of clinical attachment level in millimeters calculated for periodontal sites.

CONTACTS AND LOCATIONS:
Overall Officials: Bruno CV Gurgel, Doctor, Principal Investigator — Universidade Federal do Rio Grande do Norte
Locations (1):
- Departamento de Odontologia; Universidade Federal do Rio Grande do Norte, Natal, Rio Grande do Norte, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Quirynen M, Bollen CM, Vandekerckhove BN, Dekeyser C, Papaioannou W, Eyssen H. Full- vs. partial-mouth disinfection in the treatment of periodontal infections: short-term clinical and microbiological observations. J Dent Res. 1995 Aug;74(8):1459-67. doi: 10.1177/00220345950740080501. PMID 7560400
- [Background] Lopez NJ, Smith PC, Gutierrez J. Periodontal therapy may reduce the risk of preterm low birth weight in women with periodontal disease: a randomized controlled trial. J Periodontol. 2002 Aug;73(8):911-24. doi: 10.1902/jop.2002.73.8.911. PMID 12211502
- [Derived] Almeida ML, Duarte PM, Figueira EA, Lemos JC, Nobre CMG, Miranda TS, de Vasconcelos Gurgel BC. Effects of a full-mouth disinfection protocol on the treatment of type-2 diabetic and non-diabetic subjects with mild-to-moderate periodontitis: one-year clinical outcomes. Clin Oral Investig. 2020 Jan;24(1):333-341. doi: 10.1007/s00784-019-02927-8. Epub 2019 May 17. PMID 31102044